CLINICAL TRIAL: NCT00637221
Title: An Open Label Exploratory Study to Investigate the Safety and Effects of NPL-2009 ( 50 mg - 150 mg Single Dose) on Prepulse Inhibition Tests and Continuous Performance Tasks, in Adults With Fragile X Syndrome
Brief Title: Open Label Study Investigating Safety and Efficacy of NPL2009 50 mg - 150 mg on Prepulse Inhibition Tests and Continuous Performance Tasks, Adults With Fragile X Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neuropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NPL-2009-2-FEN-001
Record Dates: First submitted 2008-03-03; First posted 2008-03-17 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Fragile X Syndrome
Keywords: Safety; Tolerability
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NPL-2009 — Single doses of either 50mg, 100 mg or 150 mg NPL-2009

SUMMARY:
This is an open label exploratory study to investigate the safety and effects of a single dose of NPL-2009(50 mg - 150 mg) on Prepulse Inhibition (PPI) Tests and Continuous Performance Tasks (CPT) in adults with Fragile X Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 to 45 years of age.
* Diagnosis of Fragile X Syndrome.
* Females must demonstrate a negative pregnancy test at screening.
* Females of child-bearing potential must be using a medically accepted means of contraception or must remain abstinent for the duration of the study.
* Each Legally Authorised Representative (LAR, usually parent or caregiver) must have a level of understanding sufficient to provide written informed consent to all required study tests and procedures.
* Each patient must consent/assent (depending on center-specific procedures) to all required study tests and procedures.
* Permitted concomitant medications must be stable for at least 6 weeks prior to enrollment. The following concomitant medications are permitted: psychostimulants, SSRIs, atypical antipsychotics, anticonvulsants which do not have liver inducing effects, clonidine.
* Each patient must be able to swallow the capsules (2, 3 or 4) to be provided in the study.

Exclusion Criteria:

* Current treatment with anticonvulsants known to induce liver enzymes e.g. depakote
* Current treatment with N-methyl-D-aspartate (NMDA) antagonists
* Current treatment with tricyclic antidepressants
* Current treatment with typical antipsychotics
* Current treatment with lithium
* Patients planning to commence cognitive behaviour therapy during the period of the study or those who have begun cognitive behavioural therapy within 6 weeks prior to enrolment.
* History of, or current cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease which may interfere with the absorption, distribution, metabolism or excretion of the study medication.
* History of, or current cerebrovascular disease or brain trauma.
* History of, or current significant endocrine disorder, e.g. hypo or hyperthyroidism.
* History of, or current malignancy.
* Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, as assessed by the Investigator.
* Current major depressive disorder (patients must be free of the disorder for 3 months prior to enrolment).
* Judged clinically to be at risk of suicide (suicidal ideation, severe depression, or other factors), as assessed by the Investigator.
* Tourette's Disorder.
* Female patients who are either pregnant or nursing.
* Current drug abuse or dependence disorder or dependency in the 3 months prior to enrolment.
* Clinically significant abnormalities in safety laboratory tests, vital signs or EKG, as measured at screening
* Patients with significant hearing and/or visual impairments that may affect their ability to complete the test procedures
* Enrollment in another clinical trial within the previous 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for the study is that of safety and subjects will be assessed post-dose at at least hourly intervals for any signs of Adverse Events - up to allowing discharge from the unit at 6 hours post-dose | 7 Days

SECONDARY OUTCOMES:
Tolerability | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mike Snape, PhD, Study Director — Neuropharm Ltd
Locations (2):
- United States (2):
  - MIND Institute, Sacramento, California
  - Rush University Medical Centre, Chicago, Illinois